CLINICAL TRIAL: NCT04997759
Title: The Comparative Efficacy and Safety of Sugammadex and Neostigmine in Reversing Neuromuscular Blockade After General Anesthesia: A Prospective Randomized Control Study
Brief Title: Comparative Efficacy and Safety of Sugammadex and Neostigmine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202100679A3
Record Dates: First submitted 2021-07-29; First posted 2021-08-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-07

CONDITIONS: Sugammadex
Keywords: Neostigmine
MeSH Terms: interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine group (Experimental): This group will administered neostigmine for reverse the efficacy of neuromuscular blocking agent and stabilize the patient's vital signs.
  Interventions: Drug: Neostigmine and Sugammadex
- Sugammadex group (Experimental): This group will administered Sugammadex for reverse the efficacy of neuromuscular blocking agent and stabilize the patient's vital signs.
  Interventions: Drug: Neostigmine and Sugammadex

INTERVENTIONS:
Drug: Neostigmine and Sugammadex — Compare both groups efficacy of reverse the neuromuscular blocking agent

SUMMARY:
Along with unconsciousness and analgesia, use a muscle relaxant (Neuromuscular blocking agent NMBA) is now part of the classic triad of anesthesia. In surgery or interventional procedure under general anesthesia, NMBA is needed to relax the muscles of the whole body. Its purpose is to assist the placement of the endotracheal tube, avoid the participant's injury due to involuntary movements, and also enables the surgeon to have a better surgical vision, etc. Once the operation or procedure is completed, anesthesiologist will reverse the NMBA and participants are recovered from general anesthesia. It is crucial to maintain hemodynamic stability during this period. The participant's vital signs are unstable during this period because the participant is gradually recovered from anesthesia and they feel throat discomfort from endotracheal tube. Immediate extubation is encouraged in the operating theatre and full recovery of neuromuscular function must be achieved prior to extubation of the endotrachea tube.

Traditionally, acetylcholinesterase inhibitor (AChEI, such as neostigmine, pyridostigmine, edrophonium) is used to reverse the efficacy of NMBA and stabilize the participants's vital signs. However, the reversal of acetylcholine ester inhibitors is slow, the curative effect has a ceiling effect, and the need to use anticholinergics (anticholinergics) to reduce the incidence of adverse reactions and other issues. In addition, traditional muscle relaxants may also cause complications, such as postoperative residual curarization (PORC). PORC is associated with weakness of upper airway muscles and increased risk of hypoventilation and hypoxemia, as well as risk for aspiration and postoperative pulmonary complications.

Sugammadex is a new selective relaxant-binding agent that quickly and effectively reverses the effects of steroidal NMBAs, especially rocuronium and vecuronium. Compared with neostigmine, sugammadex more substantially reduces PORC, but its effects on postoperative complications require further investigation. Therefore, this study aimed to compare the effects of sugammadex and neostigmine during emergence and extubation after general anesthesia in non-cardiac surgery and interventional procedure.

DETAILED DESCRIPTION:
Investigators will include 100 participants for both groups(Suggammadex and Neostigmine) During anesthesia induction, the same drugs will be administered intravenously (propofol, fentanyl, lidocaine and rocuronium). Rocuronium, a muscle relaxant,is part of the classic triad of anesthesia. In surgery or interventional procedure under general anesthesia, NMBA is needed to relax the muscles of the whole body. Its purpose is to assist the placement of the endotracheal tube, avoid the participants injury due to involuntary movements, and also enables the surgeon to have a better surgical vision, etc. Once the operation or procedure is completed, Investigators will reverse the NMBA and participants are recovered from general anesthesia. Group A will be administered acetylcholinesterase inhibitor (AChEI, such as neostigmine, pyridostigmine, edrophonium), AChEI is used to reverse the efficacy of NMBA and stabilize the participants's vital signs. Group B will be administered sugammadex, a new selective relaxant-binding agent that quickly and effectively reverses the effects of steroidal NMBAs. Both drug should given on the time of train of four[TOF] count 4. Investigators will collect the data include: Blood pressure(extubation, one minute, two minutes and five minutes and ten minutes after), Heart rate, Saturation, extubation time and BIS.

ELIGIBILITY:
Inclusion Criteria:

* Age>20year-old
* Go Intervention or operation under general anesthesia

Exclusion Criteria:

* Chronic kidney disease(GFR<30 mL/min)
* Allergy to Sugammade/Neostigmine
* Cant extubate on the day of operation/intervention
* Neuromuscular disease
* Difficult airway
* Heart operation

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Extubation time | Since administer neostigmine or sugammadex to 30mins after Extubation
  Compare both group of extubation time and administer neostigmine or sugammadex
Blood pressure variability(systolic , diastolic and mean blood pressure) | Since administer neostigmine or sugammadex to 30mins after Extubation
  Compare both group of blood pressure variability and administer neostigmine or sugammadex
Heart rate variability | Since administer neostigmine or sugammadex to 30mins after Extubation
  Compare both group of heart rate variability and administer neostigmine or sugammadex

CONTACTS AND LOCATIONS:
Locations (1):
- Yu-Hsun-Tsai, Taoyuan District, Taiwan